CLINICAL TRIAL: NCT05052008
Title: Management of Migraine Using Enerumab and Traditional Therapy at the Time of COVID-19
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Marwa Kamal, Principle investigator, Fayoum University
Other Study IDs: Erenumab in migraine
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Migraine Disorders
Keywords: migraine, erenumab,
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Erenumab — Erenumab is monoclonal antibody used for management of migraine

SUMMARY:
The objective of this study was to assess the efficacy of erenumab on frequency of monthly migraine days in adults at baseline, 3 months and 6 months, disability in patients with chronic migraine and on post covid migraine severity

DETAILED DESCRIPTION:
Migraine is a debilitating disorder that affects 37 million people in the United States. Recently, three new injectables calcitonin gene-related peptide (CGRP) receptor antagonists-erenumab, fremanezumab, and galcanezumab-were FDA approved for prophylactic treatment of migraine in adults, that plays a key role in migraine pathophysiology. By blocking the receptor function of CGRP, these agents can reduce the total number of headache days per month and limit the need for using multiple medications. In clinical trials, these agents, which have no drug interactions and minimal adverse reactions, reduced headache days per month by as much as 50% in patients experiencing multiple migraine days each month. These new biologics, however, are more expensive for the patient compared with other prophylactic treatments

The rational of this study was to assess the efficacy of erenumab on frequency of monthly migraine days in adults at baseline, 3 months and 6 months, disability in patients with chronic migraine and on post covid migraine severity

ELIGIBILITY:
Inclusion Criteria:

* -Ages Eligible for Study: 18 Years to 65 Years (Adult, Older Adult)
* Sexes Eligible for Study: All
* History of at least 5 attacks of migraine

  -≥ 15 headache days of which ≥ 8 headache days meet criteria as migraine days during the baseline period
* chronic migraineurs with failure to more than 2 preventive treatments
* chronic migraineurs without any preventive treatments
* Naive to anti CGRP monclonal antibodies

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  • unable to understand the study requirements, the informed consent, or complete headache records as required per protocol;
* History of cluster or hemiplegic headache
* Evidence of seizure or major psychiatric disorder Cardiac or active hepatic disease
* pregnant, actively trying to become pregnant, or breast-feeding;
* episodic migraineurs,
* Other headache types
* allergy to latex;
* received nerve blocks or trigger point injections in the previous 8 weeks or plans to receive them during the study;
* prior exposure in the last 6 months to biologics or drugs specifically targeting the calcitonin gene-related peptide (CGRP) pathway;
* a psychiatric condition, that may affect the interpretation of efficacy and safety data or contraindicates the participant's participation in the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Migraine prevention is an area of a large unmet medical need, with existing prophylactic therapies often having modest efficacy and poor tolerability. Calcitonin gene-related peptide (CGRP) receptor antagonism is a novel approach to migraine preventive therapy. Erenumab is a human monoclonal antibody against CGRP receptor. The present study is a phase 3 trial intended to assess the efficacy and safety of erenumab for prevention of migraine in Egyptian adults with chronic migraine (CM).
  The study consists of a screening period (up to 24 weeks, including at baseline period), a 12-week period and a 24-week period ,.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
mean number of migraine days | 6 months
  The primary end point was the change from baseline to months 4 through 6 in the mean number of migraine days per month.
changes on migraine severity during COVID-19 infection | during the 6 months
  measuring the severity of migraine attacks on a numerical scale

SECONDARY OUTCOMES:
reduction in migraine days | during the 6 months
  Secondary end points were a 50% or greater reduction in mean migraine days per month
rate of using migraine medications | during the 6 months
  change in the number of days of use of acute migraine-specific medication
assessment of migraine effect on physical activity | during the 6 months
  change in scores on the physical-impairment and everyday-activities domains of the Migraine Physical Function Impact Diary (scale transformed to 0 to 100, with higher score

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Kamal Ahmed Tolba, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoenen J, Manise M, Nonis R, Gerard P, Timmermans G. Monoclonal antibodies blocking CGRP transmission: An update on their added value in migraine prevention. Rev Neurol (Paris). 2020 Dec;176(10):788-803. doi: 10.1016/j.neurol.2020.04.027. Epub 2020 Aug 2. PMID 32758365
- [Result] Garland SG, Smith SM, Gums JG. Erenumab: A First-in-Class Monoclonal Antibody for Migraine Prevention. Ann Pharmacother. 2019 Sep;53(9):933-939. doi: 10.1177/1060028019835166. Epub 2019 Feb 27. PMID 30813769